CLINICAL TRIAL: NCT05880706
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 for Injection and BL-B01D1 in Combination With Osimertinib Mesylate Tablets in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of BL-B01D1 and BL-B01D1 in Combination With Osimertinib Mesylate Tablets in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-203
Record Dates: First submitted 2023-05-17; First posted 2023-05-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 and BL-B01D1 in combination with Osimertinib Mesylate Tablets in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: Osimertinib Mesylate Tablets — Osimertinib Mesylate Tablets will be administered at a fixed dose of 80mg daily.

SUMMARY:
A Phase II clinical study to evaluate the efficacy and safety of BL-B01D1 for injection and BL-B01D1 in combination with Osimertinib Mesylate Tablets in patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age ≥18 years old;
4. Expected survival time ≥3 months;
5. Patients with locally advanced or metastatic non-small cell lung cancer confirmed by histopathology and/or cytology;
6. Consent to provide an archived tumor tissue sample or fresh tissue sample from the primary or metastatic site within 6 months for biomarker testing;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG ≤1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. The level of organ function must meet the requirements on the premise that no blood transfusion and no use of any cell growth factor drugs are allowed within 14 days before the screening period;
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. Fertile female subjects, or male subjects with fertile partners, must use highly effective contraception from 7 days before the first dose until 6 months after the first dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Patients with previous systemic therapy;
2. Cohort_B and Cohort_C were previously treated with EGFR-TKI;
3. Who had participated in any other clinical trial within 4 weeks before the study dose;
4. Received chemotherapy, radiotherapy, biological therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first use of study drugs;
5. Had undergone major surgery within 4 weeks before the first dose;
6. History of severe heart disease and cerebrovascular disease;
7. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
8. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
9. Current interstitial lung disease, drug-induced interstitial pneumonia, radiation pneumonitis requiring steroid therapy, or a history of these diseases;
10. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
11. Severe systemic infection within 4 weeks before screening;
12. Patients at risk for active autoimmune disease or with a history of autoimmune disease;
13. Complicated with other malignant tumors within 5 years before the first dose of medication;
14. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
15. Hypertension poorly controlled by two antihypertensive drugs;
16. Patients with poor glycemic control;
17. Patients with massive effusions, or effusions with obvious symptoms, or poorly controlled effusions;
18. Patients with active central nervous system metastases;
19. Imaging examination showed that the tumor had invaded or enveloped the large blood vessels in the abdomen, chest, neck, and pharynx;
20. Serious unhealed wound, ulcer or fracture within 4 weeks before signing the informed consent;
21. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
22. Previous history of allogeneic stem cell, bone marrow or organ transplantation;
23. Patients with a history of allergy to recombinant humanized antibody or to any of the excipients of BL-B01D1;
24. Had a history of severe neurological or psychiatric disorders;
25. Had a history of autologous or allogeneic stem cell transplantation;
26. Pregnant or lactating women;
27. Subjects scheduled for vaccination or who received live vaccine within 28 days before study randomization;
28. Other conditions for participation in the trial were not considered appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No